CLINICAL TRIAL: NCT02611492
Title: A Phase III Study, Randomized, to Evaluate the Reduction of Chemotherapy Intensity in Association With Nilotinib (Tasigna®) in Philadelphia Chromosome-positive (Ph+) ALL of Young Adults (18-59 Years Old) (GRAAPH-2014)
Brief Title: A Phase III Randomized Trial of the Reduction of Chemotherapy in Philadelphia Chromosome-positive ALL of Young Adults
Acronym: GRAAPH2014
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOM12629_1
Record Dates: First submitted 2015-11-19; First posted 2015-11-20 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-09

CONDITIONS: Philadelphia Chromosome Positive Adult Acute Lymphoblastic Leukemia
MeSH Terms: interventions — nilotinib; Methotrexate; Cytarabine; Granulocyte Colony-Stimulating Factor; Dexamethasone; Vincristine; Imatinib Mesylate; Mercaptopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Arm (A) (Active Comparator): 4 cycles + 2 interphases +Hematopoietic Stem Cell Transplantation (SCT)
  + Post-SCT Maintenance
  Interventions: Drug: Nilotinib; Drug: Methotrexate; Drug: Aracytine (Ara C); Drug: Granulocyte Colony-Stimulating Factor (G-CSF); Drug: Depomedrol; Drug: Dexamethasone; Drug: Vincristine; Drug: Imatinib; Drug: 6 Mercaptopurine (6MP)
- Light Arm (B) (Experimental): 4 cycles + 2 interphases +Hematopoietic Stem Cell Transplantation (SCT)
  + Post-SCT Maintenance
  Interventions: Drug: Nilotinib; Drug: Methotrexate; Drug: Granulocyte Colony-Stimulating Factor (G-CSF); Drug: Depomedrol; Drug: Dexamethasone; Drug: Vincristine; Drug: Imatinib; Drug: 6 Mercaptopurine (6MP)

INTERVENTIONS:
Drug: Nilotinib — 400 mg/12h per os D1 to D28 cycles 1-4 300 mg/12h per os D1-D14 interphase
Drug: Methotrexate — 1 g/m2 continuous Intravenous Infusion (CIV) D1 cycles 2 and 4 25 mg/m2 per os D1, D8 interphase
Drug: Aracytine (Ara C) — Age<45 years: 3 mg/m2/12h D2, D3 cycles 2 and 4 Age>=45 years: 1.5 mg/m2/12h D2, D3 cycles 2 and 4
  Arms: Intensive Arm (A)
Drug: Granulocyte Colony-Stimulating Factor (G-CSF) — 5µg/kg/d (SC) D6 until neutrophils > 1 G/L D15 cycles 1 and 3; D6 cycles 2 and 4
Drug: Depomedrol — 40 mg + methotrexate 15 mg + Aracytine (AraC) 40mg IT cycle 1: D1, D8, D15 IT cycles 2 and 4: D9 IT cycle 3: D1
Drug: Dexamethasone — 40 mg per os, D1-D2, D8-D9, D15-D16, D22-D23, cycles 1 and 3
Drug: Vincristine — 2 mg total dose IV, D1 D8 D15 D22 cycles 1 and 3
Drug: Imatinib — 300 mg/12h per os in post-SCT maintenance therapy for during at least 2 years
Drug: 6 Mercaptopurine (6MP) — 60 mg/m2 per os, D1 to D14, interphase

SUMMARY:
The Primary objective is to assess the non-inferiority of the experimental arm (arm B) compared to the control arm (arm A) in terms of Major Molecular Response (MMolR) after the 4th cycle (MRD4) in patients aged 18-59 years old with de novo Philadelphia positive (Ph+) acute lymphoblastic leukemia (ALL)

ELIGIBILITY:
Inclusion Criteria:

Patient

1. Whose blood and bone marrow explorations have been completed before the steroids prephase
2. Aged 18-59 years old with newly-diagnosed non previously treated Ph+ ALL according to WHO 2008 criteria (confirmed diagnosis of the Philadelphia chromosome defined by the reciprocal translocation of chromosomes 9 and 22, t(9;22) and/or presence of the BCR-ABL molecular maker)
3. With ≥ 20% bone marrow blasts
4. With Eastern Cooperative Oncology Group (ECOG) Performans Status ≤ 3
5. With or without central nervous system (CNS) or testis involvement
6. Without evolving cancer (except basal cell carcinoma of the skin or "in situ" carcinoma of the cervix) or its chemo- or radio-therapy should be finished at least since 6 months.
7. Having received no previous treatment for this hematological disease (including IT injection)
8. Having signed written informed consent
9. With efficient contraception for women of childbearing age (excluding estrogens and IUD)
10. With health insurance coverage
11. Who have received (or being receiving) the recommended steroid prephase.

Note 1: Secondary ALL (antecedent of chemo- or radio-therapy) can be included Note 2: In case of high vascular risk (see section "study management") the patient will not be able to receive nilotinib unless an ultra sound Doppler of the neck and lower limbs has been performed during the pre-phase and treatment validated by the medical coordinators of the protocol via the secretariat.

Exclusion Criteria:

Patient:

1. Previously treated with Tyrosine Kinase Inhibitor (TKI)
2. With another active malignancy
3. With general or visceral contra-indication to intensive therapy (except if considered related to the ALL):

   1. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2.5 x upper limit of normal range (ULN)
   2. Total bilirubin > 1.5 x ULN
   3. Creatinine > 1.5 x ULN or creatinine clearance <50 mL/mn
   4. Serum amylase or lipase > 1.5 x ULN or antecedents of acute pancreatitis
4. With heart failure, including at least one of the following criteria:

   1. Left ventricular ejection fraction (LVEF) <50% or below the lowest normal threshold, as determined by ECG or heart failure (NYHA grade III or IV)
   2. Impossibility to measure the QT interval on ECG
   3. Complete left bundle branch block
   4. Pacemaker
   5. Congenital long QT syndrome of known familial antecedents of long QT syndrome
   6. Antecedents or current ventricular or atrial tachyarrhythmia, clinically significant
   7. Baseline bradycardia (<50 bpm) clinically significant
   8. Corrected QT interval (QTc)> 450 msec established on the mean of 3 baseline ECG
   9. Antecedents of myocardial infarct in the past 6 months
   10. Instable angor within the past 12 months
   11. Any heart condition clinically significant (i.e. congestive heart failure, uncontrolled hypertension)
5. Active uncontrolled infection, any other concurrent disease deemed to interfere with the conduct of the study as judged by the investigator
6. Severe evolving infection, or known HIV or Human T-Lymphotropic Virus type I (HTLV1) seropositivity, or active infection by hepatitis B or C virus
7. Pregnant (beta-HCG) or nursing woman
8. Women of childbearing potential not willing to use an effective form of contraception during participation in the study and at least three months thereafter. Patient not willing to ensure not to beget a child during participation in the study and at least three months thereafter.
9. Having received an investigational treatment or participation in another trial within 30 days prior to entering this study.
10. Not able to bear with the procedures or the frequency of visits planned in the trial.
11. Unable to consent, under tutelage or curators, or judiciary safeguard

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 265 (Estimated)
Dates: Start 2016-04; Primary Completion 2020-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Major Molecular Response (MMolR) | 4 cycles (4 months)
  defined as a breakpoint cluster region (BCR)-Abelson (ABL) ratio < 0.1% in the bone marrow sample of MRD4

SECONDARY OUTCOMES:
Complete remission after cycle 1 | day 28
Cumulative incidence of treatment- and transplantation-related mortality | 2 years
Cumulative incidence of relapse | 10 years
Relapse free survival | 10 years
Event-free survival | 10 years
overall survival | 10 years
T315I mutation | 10 years
  mutations will be assessed by Reverse transcription Quantitative Polymerase Chain Reaction (RQ-PCR) sequencing in case of progression or relapse
Toxicity | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Saint Louis, Paris, France

REFERENCES:
- [Derived] Chalandon Y, Rousselot P, Chevret S, Cayuela JM, Kim R, Huguet F, Chevallier P, Graux C, Thiebaut-Bertrand A, Chantepie S, Thomas X, Vincent L, Berthon C, Hicheri Y, Raffoux E, Escoffre-Barbe M, Plantier I, Joris M, Turlure P, Pasquier F, Belhabri A, Guepin GR, Blum S, Gregor M, Lafage-Pochitaloff M, Quessada J, Lheritier V, Clappier E, Boissel N, Dombret H. Nilotinib with or without cytarabine for Philadelphia-positive acute lymphoblastic leukemia. Blood. 2024 Jun 6;143(23):2363-2372. doi: 10.1182/blood.2023023502. PMID 38452207